CLINICAL TRIAL: NCT06529653
Title: Ridge Splitting Using Autogenous Bone Wedge Versus the Conventional Intercortical Augmentation Technique in Horizontally Deficient Anterior Maxilla A Randomized Clinical Trial
Brief Title: Ridge Splitting Using Autogenous Bone Wedge Versus the Conventional Intercortical Augmentation Technique in Horizontally Deficient Anterior Maxilla
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel Salam Ibrahim Omara, masiomara, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ridge splitting
Record Dates: First submitted 2024-07-24; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Horizontal Ridge Deficiency
Keywords: ridge splitting, bone wedge, mixed bone particles, horizontally deficient ridge, aesthetic zone, ridge augmentation.

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Other): the group using an autogenous bone wedge harvested from the chin interpositioned between split cortices in the anterior maxilla to manage the horizontal deficiency of the ridge.
  Interventions: Procedure: autogenous bone wedge
- control group (Other): the group used mixed autogenic and xenogenic bone particles that interposed between split cortices in anterior maxilla to manage the horizontal deficiency of the ridge
  Interventions: Procedure: autogenous bone wedge

INTERVENTIONS:
Procedure: autogenous bone wedge — autogenous bone block harvested from chin and adjusted to be wedged intercortical in split ridge

SUMMARY:
The current study aimed to evaluate both the quality and quantity of gained and maintained bone width after ridge splitting utilizing autogenic bone wedges versus mixed bone particles for horizontal ridge augmentation in the anterior esthetic zone.

DETAILED DESCRIPTION:
This randomized clinical study included 20 patients with a horizontally deficient ridge in the esthetic region. Two groups were divided according to the type of intercortical bone graft used after ridge splitting: 10 patients for each. (The intervention group) had grafting with autogenous bone wedges harvested from the chin, and (the control group) had mixed (autogenic and xenogenic) bone particles.

ELIGIBILITY:
Inclusion Criteria:

1. All patients possessed partially edentulous anterior maxillary ridge with the following criteria

   1. The anterior maxillary vertical dimension was more than ten mm measured from the alveolar crest to the basal bone of the maxilla.
   2. The horizontal alveolar dimension varies from 3-5 mm at the crest and 6-8 mm at the basal part of the ridge measured from the labial cortex to the lingual cortex.
2. All patients were free from any medical conditions that may affect bone healing .
3. No local pathosis that may interfere with bone healing.
4. No previous grafting procedures at the indicated edentulous ridge.

   -

   Exclusion Criteria:

1- Patients suffering from any systemic disease that may affect bone healing. 2- Patients with less than 3mm labio palatal alveolar ridge width. 3- Ridge with inadequate vertical bone height. 4- Presence of any local pathosis that may interfere with bone healing. 5- Patients unable to continue the whole follow up.

-

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
bone width in (mm) by cone beam pre, immediate post operative and 6 months postoperative | 6 months
  after ridge augmentation in both groups, the bone width will be measured immediately postoperatively and 6 months postoperatively with cone beam and the measurements of the three intervals (pre-, immediate and 6 months postoperatively) will be compared in both groups to evaluate the amount of gained and maintained bone width

SECONDARY OUTCOMES:
percentage of areas of new bone (%) | 6 months
  The harvested core biopsies would be stained with H&E and Massons trichrome stain and be microscopically examined to determine percentage areas of newly formed bone

CONTACTS AND LOCATIONS:
Locations (1):
- oral and maxillo facial Surgery Department; Faculty of dentistry, Cairo University., Cairo, Egypt

REFERENCES:
- [Background] Atef M, Osman AH, Hakam M. Autogenous interpositional block graft vs onlay graft for horizontal ridge augmentation in the mandible. Clin Implant Dent Relat Res. 2019 Aug;21(4):678-685. doi: 10.1111/cid.12809. Epub 2019 Jul 1. PMID 31260166
- [Derived] Omara M, Mekhemer S, Mansour S, Ahmed Y. Ridge splitting using autogenous bone wedge versus the conventional intercortical augmentation technique in horizontally deficient anterior maxilla: a randomized clinical trial. BMC Oral Health. 2025 Jun 21;25(1):955. doi: 10.1186/s12903-025-06345-z. PMID 40544250
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31260166/